CLINICAL TRIAL: NCT00483782
Title: ICON7 - A Randomised, Two-Arm, Multi-Centre Gynaecologic Cancer InterGroup Trial of Adding Bevacizumab to Standard Chemotherapy (Carboplatin and Paclitaxel) in Patients With Epithelial Ovarian Cancer
Brief Title: Carboplatin and Paclitaxel With or Without Bevacizumab in Treating Patients With Newly Diagnosed Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: MREC-ICON7; CDR0000548777 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2005-003929-22; ISRCTN91273375; ROCHE-MREC-ICON7; EU-20730; MREC-06/MRE02/52
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2012-04

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage IV ovarian epithelial cancer; Brenner tumor; ovarian carcinosarcoma; ovarian clear cell cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian mucinous cystadenocarcinoma; ovarian serous cystadenocarcinoma; ovarian undifferentiated adenocarcinoma; stage IA ovarian epithelial cancer; stage IB ovarian epithelial cancer; stage IC ovarian epithelial cancer; stage IIA ovarian epithelial cancer; stage IIB ovarian epithelial cancer; stage IIC ovarian epithelial cancer; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; stage IA fallopian tube cancer; stage IB fallopian tube cancer; stage IC fallopian tube cancer; stage IIA fallopian tube cancer; stage IIB fallopian tube cancer; stage IIC fallopian tube cancer; stage IIIA fallopian tube cancer; stage IIIB fallopian tube cancer; stage IIIC fallopian tube cancer; stage IV fallopian tube cancer; stage IA primary peritoneal cavity cancer; stage IB primary peritoneal cavity cancer; stage IC primary peritoneal cavity cancer; stage IIA primary peritoneal cavity cancer; stage IIB primary peritoneal cavity cancer; stage IIC primary peritoneal cavity cancer; stage IIIA primary peritoneal cavity cancer; stage IIIB primary peritoneal cavity cancer; stage IIIC primary peritoneal cavity cancer; stage IV primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — Bevacizumab; Carboplatin; Paclitaxel

INTERVENTIONS:
Biological: bevacizumab
Drug: carboplatin
Drug: paclitaxel
Other: questionnaire administration
Other: study of socioeconomic and demographic variables
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. It is not yet known whether giving carboplatin and paclitaxel together with bevacizumab is more effective than carboplatin and paclitaxel alone in treating patients with ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cavity cancer.

PURPOSE: This randomized phase III trial is studying carboplatin, paclitaxel, and bevacizumab to see how well they work compared with carboplatin and paclitaxel alone in treating patients with newly diagnosed ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the progression-free survival and overall survival of patients with newly diagnosed ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer treated with carboplatin and paclitaxel with vs without bevacizumab.

Secondary

* Compare the response rate in patients treated with these regimens.
* Compare the duration of tumor response in patients treated with these regimens.
* Compare the biological progression-free interval, as measured by increasing CA 125 levels, in patients treated with these regimens.
* Compare the safety (e.g., adverse events, laboratory results, and performance status) of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.
* Compare the cost-effectiveness of these regimens in these patients.

OUTLINE: This is a multicenter, open-label, randomized, controlled study. Patients are stratified according to FIGO stage (stage I-III with residual disease ≤ 1 cm vs stage I-III with residual disease > 1 cm vs stage IV disease), intended time to start chemotherapy after surgery (≤ 4 weeks vs > 4 weeks), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I (control): Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive bevacizumab IV over 30-90 minutes followed by paclitaxel IV over 3 hours and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients then continue to receive bevacizumab alone every 3 weeks for 12 courses.

Quality of life is assessed at baseline, before every course, every 6 weeks for 1 year, every 3 months until disease progression or for up to 2 years, and then at 3 years. Health economic data is assessed periodically, including days of inpatient hospitalization visits, outpatient visits, and use of anticancer therapies.

After completion of study treatment, patients are followed every 3-6 months for 5 years and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer

  * Newly diagnosed disease
* Meets 1 of the following staging criteria:

  * High-risk stage I or IIA disease (grade 3 disease or clear cell carcinoma only)
  * Stage IIB-IV disease (all grades and all histological types)
* Must have undergone initial surgery (e.g., debulking cytoreductive surgery or a biopsy if the patient has stage IV disease) within the past 6 weeks

  * Patients with stage IV disease for which initial surgical debulking was not appropriate are eligible provided the following criteria are met:

    * Stage IV disease diagnosed by histology
    * No planned surgery prior to disease progression, including interval debulking surgery
* Patients with prior early-stage ovarian epithelial or fallopian tube carcinoma treated with surgery alone are eligible at the time of diagnosis of abdominopelvic recurrence provided no further interval cytoreductive therapy is planned prior to disease progression
* Synchronous primary endometrial carcinoma or a past history of primary endometrial carcinoma allowed provided the following criteria are met:

  * Disease ≤ stage IB
  * No more than superficial myometrial invasion
  * No lymphovascular invasion
  * Not poorly differentiated (i.e., no grade 3, papillary serous, or clear cell disease)
* Measurable or nonmeasurable disease
* No ovarian nonepithelial cancer, including malignant mixed Müllerian tumors
* No borderline tumors (e.g., tumors of low malignant potential)
* No history or clinical suspicion of brain metastases or spinal cord compression

  * CT scan or MRI of the brain is mandatory (within 4 weeks prior to randomization) in case of suspected brain metastases
  * Spinal MRI is mandatory (within 4 weeks prior to randomization) in case of suspected spinal cord compression

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 12 weeks
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL (can be post-transfusion)
* INR ≤ 1.5
* APTT ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* ALT and AST ≤ 2.5 times ULN
* Creatinine ≤ 2.0 mg/dL
* Proteinuria ≤ 1+ by urine dipstick OR ≤ 1 g by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 weeks after completion of study therapy
* No significant traumatic injury within the past 4 weeks
* No cerebrovascular accident, transient ischemic attack, or subarachnoid hemorrhage within the past 6 months
* No other malignancies within the past 5 years except for adequately treated carcinoma in situ of the cervix, and/or basal cell skin cancer, and/or early endometrial carcinoma
* No pre-existing sensory or motor neuropathy ≥ grade 2
* No history or evidence of CNS disease (e.g., uncontrolled seizures) by neurological examination unless adequately treated with standard medical therapy
* No history or evidence of thrombotic or hemorrhagic disorders
* No uncontrolled hypertension (i.e., blood pressure > 150/100 mm Hg despite antihypertensive therapy)
* No known hypersensitivity to bevacizumab and its excipients, chemotherapy, or Cremophor EL
* No nonhealing wound, ulcer, or bone fracture

  * Patients with granulating incisions healing by secondary intention with no evidence of facial dehiscence or infection are eligible but require three weekly wound examinations
* No clinically significant cardiovascular disease, including any of the following:

  * Myocardial infarction or unstable angina within the past 6 months
  * New York Heart Association class II-IV congestive heart failure
  * Poorly controlled cardiac arrhythmia despite medication

    * Rate-controlled atrial fibrillation allowed
  * Peripheral vascular disease ≥ grade 3 (i.e., symptomatic and interfering with activities of daily living requiring repair or revision)
* No evidence of other disease or condition, metabolic dysfunction, physical examination findings, or laboratory findings that would contraindicate the use of an investigational drug or put the patient at high-risk for treatment-related complications

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since other prior surgery or open biopsy
* No prior systemic therapy for ovarian cancer (e.g., chemotherapy, monoclonal antibody therapy, tyrosine kinase inhibitor therapy, or hormonal therapy)
* Prior adjuvant chemotherapy allowed for other malignancies (e.g., breast or colorectal carcinoma) if malignancy was diagnosed over 5 years ago with no evidence of subsequent recurrence
* No prior mouse CA 125 antibody
* No prior radiotherapy to the abdomen or pelvis
* More than 10 days since prior and no concurrent chronic use of acetylsalicylic acid (> 325 mg/day)

  * Low-dose (< 325 mg/day) acetylsalicylic acid allowed
* More than 10 days since prior and no concurrent full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes

  * Use of therapy for line patency allowed provided INR < 1.5
* More than 30 days since prior and no other concurrent investigational agent or participation in another clinical trial
* No other concurrent systemic antitumor agents
* No concurrent surgery
* No concurrent maintenance chemotherapy or intraperitoneal chemotherapy (including cytotoxic chemotherapy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1520 (Estimated)
Dates: Start 2006-04

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Duration of overall survival
Objective response rate
Duration of response
Biological progression-free interval as measured by increasing CA 125 levels
Safety as measured by NCI CTAE version 3.0
Quality of life
Health economics

CONTACTS AND LOCATIONS:
Overall Officials: Tim J. Perren, MD, Study Chair — Leeds Cancer Centre at St. James's University Hospital
Locations (142):
- Australia (16):
  - Cancer Therapy Centre at Liverpool Hospital, Liverpool, New South Wales
  - Prince of Wales Private Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Sydney Cancer Centre at Royal Prince Alfred Hospital, Sydney, New South Wales
  - Newcastle Mater Misericordiae Hospital, Waratah, New South Wales
  - Westmead Institute for Cancer Research at Westmead Hospital, Wentworthville, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - Royal Adelaide Hospital Cancer Centre, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Royal Women's Hospital, Carlton, Victoria
  - Mercy Hospital for Women, East Melbourne, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Murray Valley Private Hospital and Cancer Treatment Centre, Wodonga, Victoria
  - Sir Charles Gairdner Hospital - Perth, Perth, Western Australia
- France (29):
  - Centre Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Clinique Tivoli, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Hopital Louis Pasteur, Colmar
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Institut Prive de Cancerologie, Grenoble
  - Hopital Andre Mignot, Le Chesnay
  - Centre Jean Bernard, Le Mans
  - Centre Leon Berard, Lyon
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre D'Oncologie De Gentilly, Nancy
  - Centre Catherine de Sienne, Nantes
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Hopital Europeen Georges Pompidou, Paris
  - Institut Curie Hopital, Paris
  - Hotel Dieu de Paris, Paris
  - Hopital Cochin, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Centre Rene Huguenin, Saint-Cloud
  - Hopital Universitaire Hautepierre, Strasbourg
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
- Germany (50):
  - Evang. Waldkrankenhaus Spandau, Berlin
  - Charite University Hospital - Campus Virchow Klinikum, Berlin
  - Klinikum Bremen-Mitte, Bremen
  - Praxis Dres. F.& G. Doering, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Kreiskrankenhaus, Ebersberg
  - Universitaetsklinikum Essen, Essen
  - Elisabeth-Krankenhaus, Essen
  - Staedtische Kliniken Esslingen, Esslingen am Neckar
  - Onkologie Bethanien, Frankfurt
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Staedtische Kliniken Frankfurt am Main - Hoechst, Frankfurt
  - Universitaetsfrauenklinik Freiburg, Freiburg im Breisgau
  - Franziskus Hospital Hardenberg, Georgsmarienhütte
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Universitaetsklinikum Halle, Halle
  - Henriettenstiftung Frauenklinik, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - St. Vincentius - Kliniken, Karlsruhe
  - Klinikum Kassel, Kassel
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Kreiskrankenhaus Lahr, Lahr
  - Kreiskrankenhaus Leonberg - Frauenklinik, Leonberg
  - Asklepios Klinik Lich, Lich
  - St. Vincenz Hospital Limburg, Limburg
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck
  - Staedtisches Klinikum Lueneburg, Lüneburg
  - Klinik St. Marienstift Magdeburg, Magdeburg
  - St. Vincenz und Elisabeth Hospital, Mainz
  - Universitaetsklinikum Giessen und Marburg GmbH - Marburg, Marburg
  - Klinikum Minden, Minden
  - I. Frauenklinik und Hebammenschule der Ludwig-Maximillians Universitaet Muenchen, Munich
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Staedtisches Klinikum Neunkirchen gGmbH, Neunkirchen
  - Lukaskrankenhaus Neuss, Neuss
  - Klinikum Offenback GmbH, Offenbach
  - Saint Vincenz-Krankenhaus Paderborn, Paderborn
  - Klinikum Dorothea Christiane Erxleben - Quedlingburg, Quedlinburg
  - Krankenhaus St. Elisabeth - Ravensburg, Ravensburg
  - St. Marien - Krankenhaus Siegen GMBH, Siegen
  - Kliniken Landkreis Sigmaringen GMBH, Sigmaringen
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Marienhospital Stuttgart, Stuttgart
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
  - Marien-Hospital Witten, Witten
  - Klinikum der Stadt Wolfsburg, Wolfsburg
  - Praxis Fuer Haemotologie Und Internistischer Onkologie, Wuppertal
- Norwegian Radium Hospital, Oslo, Norway
- United Kingdom (46):
  - North Devon District Hospital, Barnstaple, England
  - Broomfield Hospital, Broomfield, England
  - Queen's Hospital, Burton-on-Trent, England
  - Addenbrooke's Hospital, Cambridge, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Queen Elizabeth Hospital, Gateshead, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - Ipswich Hospital, Ipswich, England
  - Airedale General Hospital, Keighley, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - University College of London Hospitals, London, England
  - Guy's Hospital, London, England
  - St. George's Hospital, London, England
  - Hammersmith Hospital, London, England
  - Mid Kent Oncology Centre at Maidstone Hospital, Maidstone, England
  - Christie Hospital, Manchester, England
  - Queen Elizabeth The Queen Mother Hospital, Margate, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Northampton General Hospital, Northampton, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Nottingham City Hospital, Nottingham, England
  - Churchill Hospital, Oxford, England
  - Derriford Hospital, Plymouth, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth Hants, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - Stoke Mandeville Hospital, Shrewsbury, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - Southampton General Hospital, Southampton, England
  - Staffordshire General Hospital, Stafford, England
  - Royal Marsden - Surrey, Sutton, England
  - Great Western Hospital, Swindon, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - Yeovil District Hospital, Yeovil - Somerset, England
  - Centre for Cancer Research and Cell Biology at Queen's University Belfast, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - South West Wales Cancer Institute, Swansea, Wales

REFERENCES:
- [Background] Dhillon S. Bevacizumab combination therapy: for the first-line treatment of advanced epithelial ovarian, fallopian tube or primary peritoneal cancer. Drugs. 2012 May 7;72(7):917-30. doi: 10.2165/11208940-000000000-00000. PMID 22515620
- [Result] Perren TJ, Swart AM, Pfisterer J, Ledermann JA, Pujade-Lauraine E, Kristensen G, Carey MS, Beale P, Cervantes A, Kurzeder C, du Bois A, Sehouli J, Kimmig R, Stahle A, Collinson F, Essapen S, Gourley C, Lortholary A, Selle F, Mirza MR, Leminen A, Plante M, Stark D, Qian W, Parmar MK, Oza AM; ICON7 Investigators. A phase 3 trial of bevacizumab in ovarian cancer. N Engl J Med. 2011 Dec 29;365(26):2484-96. doi: 10.1056/NEJMoa1103799. PMID 22204725
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Vaughan S, Coward JI, Bast RC Jr, Berchuck A, Berek JS, Brenton JD, Coukos G, Crum CC, Drapkin R, Etemadmoghadam D, Friedlander M, Gabra H, Kaye SB, Lord CJ, Lengyel E, Levine DA, McNeish IA, Menon U, Mills GB, Nephew KP, Oza AM, Sood AK, Stronach EA, Walczak H, Bowtell DD, Balkwill FR. Rethinking ovarian cancer: recommendations for improving outcomes. Nat Rev Cancer. 2011 Sep 23;11(10):719-25. doi: 10.1038/nrc3144. PMID 21941283